CLINICAL TRIAL: NCT03601429
Title: Dietary Supplementation of Lactogyn in Women With Bacterial Vaginosis: a Randomized Clinical Trial
Brief Title: Dietary Supplementation of Lactogyn in Women With Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vesale Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BV-SVG-A001
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactogyn (Experimental): 1 capsule of Lactogyn 2 times daily for the first 7 days then 1 time daily for 4 months
  Interventions: Dietary Supplement: Lactogyn
- Placebo (Placebo Comparator): 1 capsule of Placebo Comparator 2 times daily for the first 7 days then 1 time daily for 4 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactogyn — capsules
  Arms: Lactogyn
Dietary Supplement: Placebo — capsules
  Arms: Placebo

SUMMARY:
The objective of the study is to determine clinical efficacy of Lactogyn (Lactobacillus Crispatus, L. brevis, L.acidophilus) in prevention of recurrent BV

DETAILED DESCRIPTION:
According to classification, this is a phase 2 randomized parallel group prospective controlled dietary study to evaluate efficacy of a dietary supplement, a combination of L. crispatus LMG S-29995, L. brevis, and L. acidophilus in women aged from 18 through 45 years suffering from rBV. The 2 phase of the study has been ascribed as there is no evidence that oral capsules with L. crispatus LMG S-29995, L. brevis, and L. acidophilus have a potential efficacy in rBV.

Qualifying women received a combination of the three probiotic strains with a half daily recommended dose of vitamin C or just vitamin C without probiotics, a control supplementation, via oral route of administration for up to 120 days. During the intake of active or control formulations, participants kept a structured 120-DSD, where they recorded test capsules intake, screen for symptoms of bacterial vaginosis, and food intolerance events.

Based on repeat physical examination with application of Amsel and Nugent criteria the main conclusions over the efficacy of probiotic strains were made.

ELIGIBILITY:
Inclusion criteria

1. Informed consent form signed;
2. Age: 18-45 years;
3. Able to swallow capsules;
4. Recent symptomatic BV successfully treated with metronidazole tablets in a dose of 500 mg 2 times daily for 7 days;
5. Less than 48 hours after treatment of acute BV defined as three out of four Amsel criteria;
6. Willing to communicate intimate history for the study purposes;
7. Consent not to use spermicides for 4 months after starting TDC;
8. Stated availability throughout the study period and a mobile phone.

Exclusion criteria

1. Post-menopausal;
2. Pregnancy or high risk of;
3. Breast feeding;
4. Currently active STD as determined by history, physical examination, and laboratory tests;
5. Diabetes mellitus;
6. Inflammatory bowel disease;
7. Alcohol or drug addiction as guessed by investigator;
8. Absence of refrigerator;
9. Known moderate to severe disease of any systems;
10. Difficulty to comprehend study requirements as judged by physician;
11. Any erosions, herpes like lesions, cervicitis during vaginal examination;
12. Treatment of BV with other than metronidazole antibiotic;
13. Use of any investigational drug within the previous 30 days;
14. Use of drugs that suppress the immune system.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Percent change in recurrence of BV during Lactogyn supplementation | 4 months
  Percent change in recurrence of BV during the 4 months of dietary supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Karl Richir, Study Director — Vesale Pharma
Locations (1):
- Sergiy V. Gerasymov, MD, PhD, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No